CLINICAL TRIAL: NCT06483594
Title: Prediction and Prognostic Analysis of Liver Abscess Formation After Transcatheter Arterial Chemoembolization for Hepatocellular Carcinoma : a Retrospective Multicenter Nested Case-control Study (CHANCE 2407)
Brief Title: Prediction and Prognostic Analysis of Liver Abscess Formation After Transcatheter Arterial Chemoembolization for Hepatocellular Carcinoma (CHANCE 2407)
Status: Not yet recruiting | Type: Observational
Sponsor: Shengjing Hospital (Other)
Collaborators: First Hospital of China Medical University (Other); Zhongda Hospital (Other); Changzhou No.2 People's Hospital (Other); Tianjin Medical University General Hospital (Other); Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Zhihui Chang, Professor, Shengjing Hospital
Other Study IDs: 2024PS1094K
Record Dates: First submitted 2024-06-10; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: TACE; HCC - Hepatocellular Carcinoma; Liver Abscess
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Abscess

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with liver abscess formation after TACE for HCC
- Patients without liver abscess after TACE with HCC

SUMMARY:
Liver abscess is a rare but serious complication of hepatocellular carcinoma after TACE, with an incidence of less than 1% reported in previous literature. Studies have shown that history of biliary tract disease, tumor size, embolization materials and embolization endpoint selection may be related to the occurrence of abscess. In recent years, with the wide application of targeted and immune drugs, there have been reports of multiple cases of liver abscess after single target immunotherapy for liver cancer, and there have also been studies showing that TACE combined with targeted immunotherapy can significantly increase the degree of liquefaction necrosis and increase the risk of liver abscess. However, these studies are single-center reports with small sample size and low level of evidence. Therefore, it is of great clinical significance to explore the risk factors of liver abscess after TACE and build a prediction model by using multi-center and large sample data. The formation of liver abscess after TACE means a large range of tissue liquefaction necrosis. There are reports of high incidence of early recurrence and metastasis of liquefaction necrosis. Some studies also show that tumor necrosis is more complete when liver abscess is combined with complete remission. In previous studies, ORR in patients with liver cancer complicated with liver abscess ranged from 18.75%-100%, with significant differences in reports from different centers. The effect of specific abscess formation on TACE efficacy of liver cancer remains to be determined. Therefore, the second research focus of this project is to explore the effect of liver abscess formation after TACE on prognosis of liver cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Case group inclusion criteria:

   1. Time period of inclusion: 2009-2023 (15 years)
   2. Patients with HCC diagnosed by clinical or pathological criteria according to the National Health Commission guidelines for the diagnosis and treatment of primary liver cancer who underwent TACE after surgery and developed postoperative liver abscess.
   3. Appendix: Diagnostic criteria for liver abscess after TACE:

   Condition 1: CT images show typically low-density lesions with or without air and fluid levels

   Condition 2:
   * positive blood culture
   * Percutaneous drainage or aspiration is purulent or culture-positive
   * Symptoms of infection such as fever/chills, accompanied by elevated inflammatory markers such as white blood cell count, C-reactive protein, or procalcitonin.
2. Control group inclusion criteria

   1. Patients with HCC without liver abscess who underwent TACE in the same center within the week of treatment in the case group.

      -

      Exclusion Criteria:

   <!-- -->

   1. Clinical and follow-up data were incomplete
   2. Loss to follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HCC patients from hospital interventional wards receiving TACE
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-06-30 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Whether combined targeted therapy was a risk factor for liver abscess formation after TACE. | one year
  The targeted treatment of patients with and without liver abscess after TACE was collected, and conclusion was drawn by univariate and multivariate analysis.
Whether combined immunotherapy was a risk factor for liver abscess formation after TACE. | one year
  The immunotherapy of patients with and without liver abscess after TACE was collected, and conclusion was drawn by univariate and multivariate analysis.

SECONDARY OUTCOMES:
Survival time of patients with liver abscess formation after TACE. | one year
  Patients with liver abscess formation after TACE were followed up regularly to determine their survival status.

IPD SHARING:
Plan to Share IPD: No